CLINICAL TRIAL: NCT02553317
Title: A Phase III Double-blind, Randomized, Parallel Group, Multicenter Placebo-controlled Trial to Study the Efficacy and Safety of Caplacizumab in Patients With Acquired Thrombotic Thrombocytopenic Purpura
Brief Title: Phase III Trial With Caplacizumab in Patients With Acquired Thrombotic Thrombocytopenic Purpura
Acronym: HERCULES
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ablynx, a Sanofi company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALX0681-C301; 2015-001098-42 (EudraCT Number)
Record Dates: First submitted 2015-09-14; First posted 2015-09-17 (Estimated); Results first posted 2019-05-22 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2019-05

CONDITIONS: Acquired Thrombotic Thrombocytopenic Purpura
MeSH Terms: conditions — Purpura, Thrombotic Thrombocytopenic | interventions — caplacizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (2):
- Caplacizumab (Experimental): Caplacizumab 10 mg once daily
  Interventions: Biological: Caplacizumab
- Placebo (Placebo Comparator): Placebo once daily
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Caplacizumab — * First day of treatment: 10 mg intravenous (i.v.) injection prior to plasma exchange (PE) followed by a 10 mg subcutaneous (s.c.) injection (in the abdominal region) after completion of PE on that day.
  * Subsequent days of treatment during PE: daily 10 mg s.c. injection (in the abdominal region) following PE.
  * Treatment after PE period: daily 10 mg s.c. injections for 30 days. If the underlying immunological disease was not resolved, treatment could be extended for a maximum of 4 additional 1-week periods (i.e., 28 days) and was to be accompanied by optimization of immunosuppression.
  Other Names: ALX-0081
  Arms: Caplacizumab
Biological: Placebo — * First day of treatment: i.v. injection prior to PE followed by a s.c. injection (in the abdominal region) after completion of PE on that day.
  * Subsequent days of treatment during PE: daily s.c. injection (in the abdominal region) following PE.
  * Treatment after PE period: daily s.c. injections for 30 days. If the underlying immunological disease was not resolved, treatment could be extended for a maximum of 4 additional 1-week periods (i.e., 28 days) and was to be accompanied by optimization of immunosuppression.
  Other Names: ALX-0081 Placebo
  Arms: Placebo

SUMMARY:
The study was a Phase III, double-blind, placebo-controlled, randomized study to evaluate the efficacy of caplacizumab in more rapidly restoring normal platelet counts as measure of prevention of further microvascular thrombosis

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female ≥ 18 years of age at the time of signing the informed consent form (ICF).
2. Clinical diagnosis of acquired thrombotic thrombocytopenic purpura (aTTP) (initial or recurrent), which included thrombocytopenia and microscopic evidence of red blood cell fragmentation (e.g., schistocytes).
3. Required initiation of daily PE treatment and had received 1 PE treatment prior to randomization
4. Others as defined in the protocol

Exclusion Criteria:

1. Platelet count ≥100×10E9/L.
2. Serum creatinine level >200 µmol/L in case platelet count is > 30×10E9/L
3. Known other causes of thrombocytopenia
4. Congenital TTP (known at the time of study entry).
5. Pregnancy or breast-feeding.
6. Subjects who were previously enrolled in a clinical study with caplacizumab and received caplacizumab or for whom the assigned treatment arm is unknown
7. Others as defined in the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Ablynx NV
Locations (100):
- United States (18):
  - Investigator Site, Birmingham, Alabama
  - Investigator Site, Los Angeles, California
  - Investigator Site, Atlanta, Georgia
  - Investigator Site, Boston, Massachusetts
  - Investigator Site, St Louis, Missouri
  - Investigator Site, Rochester, New York
  - Investigator Site, Valhalla, New York
  - Investigator Site, Chapel Hill, North Carolina
  - Investigator Site, Durham, North Carolina
  - Investigator Site, Winston-Salem, North Carolina
  - Investigator SIte, Cleveland, Ohio
  - Investigator Site, Columbus, Ohio
  - Investigator Site, Oklahoma City, Oklahoma
  - Investigator Site, Pittsburgh, Pennsylvania
  - Investigator Site, Charleston, South Carolina
  - Investigator Site, Greenville, South Carolina
  - Investigator Site, Houston, Texas
  - Investigator Site, Salt Lake City, Utah
- Australia (9):
  - Investigator Site, Brisbane
  - Investigator Site 1, Melbourne
  - Investigator Site 2, Melbourne
  - Investigator Site 3, Melbourne
  - Investigator Site 4, Melbourne
  - Investigator Site 5, Melbourne
  - Investigator Site, Perth
  - Investigator Site 1, Sydney
  - Investigator Site 2, Sydney
- Investigator Site, Vienna, Austria
- Belgium (5):
  - Investigator Site, Antwerp
  - Investigator Site, Brussels
  - Investigator Site, Haine-Saint-Paul
  - Investigator Site, La Louvière
  - Investigator Site, Leuven
- Canada (3):
  - Invesigator Site, Montreal, Quebec
  - Investigator Site, London
  - Investigator Site, Toronto
- Czechia (4):
  - Investigator Site, Brno
  - Investigator Site, Hradec Králové
  - Investigator Site, Olomouc
  - Investigator Site, Ostrava-Poruba
- France (11):
  - Investigator Site, Caen
  - Investigator Site, Lille
  - Investigator Site, Marseille
  - Investigator Site, Nantes
  - Investigator Site 1, Paris
  - Investigator Site 2, Paris
  - Investigator Site 3, Paris
  - Investigator Site 4, Paris
  - Investigator site 5, Paris
  - Investigator Site, Rouen
  - Investigator Site, Salouël
- Germany (8):
  - Investigator site, Cologne
  - Investigator site 1, Dresden
  - Investigator site 2, Dresden
  - Investigator site, Erlangen
  - Investigator site, Göppingen
  - Investigator site, Kiel
  - Investigator site, Leipzig
  - Investigator site, Würzburg
- Hungary (3):
  - Investigator Site 1, Budapest
  - Investigator Site 2, Budapest
  - Investigator Site, Debrecen
- Israel (8):
  - Investigator Site 1, Be’er Ya‘aqov
  - Investigator Site 2, Be’er Ya‘aqov
  - Investigator Site, Haifa
  - Investigator Site 1, Jerusalem
  - Investigator Site 2, Jerusalem
  - Investigator Site, Nahariya
  - Investigator Site, Petah Tikva
  - Investigator Site, Tel Aviv
- Italy (6):
  - Investigator Site, Catania
  - Investigator Site 1, Milan
  - Investigator Site 2, Milan
  - Investigator Site, Pesaro
  - Investigator Site, Rome
  - Investigator Site, Vicenza
- Netherlands (4):
  - Investigator Site, Amersfoort
  - Investigator Site, Leiden
  - Investigator Site, Rotterdam
  - Investigator Site, Veldhoven
- Spain (7):
  - Investigator Site 1, Barcelona
  - Investigator Site 2, Barcelona
  - Investigator Site, Madrid
  - Investigator Site, Seville
  - Investigator Site 1, Valencia
  - Investigator Site 2, Valencia
  - Investigator site 3, Valencia
- Switzerland (2):
  - Investigator Site, Bern
  - Investigator Site, Zurich
- Turkey (Türkiye) (7):
  - Investigator Site, Ankara
  - Investigator Site 1, Denizli
  - Investigator Site 2, Denizli
  - Investigator site 3, Denizli
  - Investigator Site, Istanbul
  - Investigator Site, Kayseri
  - Investigator Site, Trabzon
- United Kingdom (4):
  - Investigator Site, Bristol
  - Investigator Site, Liverpool
  - Investigator Site 1, London
  - Investigator Site 2, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Peyvandi F, Cataland S, Scully M, Coppo P, Knoebl P, Kremer Hovinga JA, Metjian A, de la Rubia J, Pavenski K, Minkue Mi Edou J, De Winter H, Callewaert F. Caplacizumab prevents refractoriness and mortality in acquired thrombotic thrombocytopenic purpura: integrated analysis. Blood Adv. 2021 Apr 27;5(8):2137-2141. doi: 10.1182/bloodadvances.2020001834. PMID 33881463
- [Derived] Knoebl P, Cataland S, Peyvandi F, Coppo P, Scully M, Kremer Hovinga JA, Metjian A, de la Rubia J, Pavenski K, Minkue Mi Edou J, De Winter H, Callewaert F. Efficacy and safety of open-label caplacizumab in patients with exacerbations of acquired thrombotic thrombocytopenic purpura in the HERCULES study. J Thromb Haemost. 2020 Feb;18(2):479-484. doi: 10.1111/jth.14679. Epub 2019 Dec 9. PMID 31691462
- [Derived] Scully M, Cataland SR, Peyvandi F, Coppo P, Knobl P, Kremer Hovinga JA, Metjian A, de la Rubia J, Pavenski K, Callewaert F, Biswas D, De Winter H, Zeldin RK; HERCULES Investigators. Caplacizumab Treatment for Acquired Thrombotic Thrombocytopenic Purpura. N Engl J Med. 2019 Jan 24;380(4):335-346. doi: 10.1056/NEJMoa1806311. Epub 2019 Jan 9. PMID 30625070

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 145 subjects was randomized at 55 sites located in Europe (34 sites; 91 subjects), Asia (4 sites, 6 subjects), Australia (3 sites, 3 subjects), and North America (14 sites; 45 subjects). Consent was obtained from the first subject on 19 November 2015; the last subject completed the final visit on 16 August 2017.
Pre-assignment Details: Of the 149 subjects screened, 4 were screen failures and 145 were randomly assigned to treatment (Intent-to-treat [ITT] population). All, except 1 subject who withdrew consent, received study drug and were included in the safety population and in the modified ITT (mITT) population.
Groups:
- Caplacizumab: Caplacizumab 10 mg once daily
  Caplacizumab:
  * First day of treatment: 10 mg intravenous (i.v.) injection prior to plasma exchange (PE) followed by a 10 mg subcutaneous (s.c.) injection (in the abdominal region) after completion of PE on that day.
  * Subsequent days of treatment during PE: daily 10 mg s.c. injection (in the abdominal region) following PE.
  * Treatment after PE period: daily 10 mg s.c. injections for 30 days. If the underlying immunological disease was not resolved, treatment could be extended for a maximum of 4 additional 1-week periods (i.e., 28 days) and was to be accompanied by optimization of immunosuppression.
- Placebo: Placebo once daily
  Placebo:
  * First day of treatment: i.v. injection prior to PE followed by a s.c. injection (in the abdominal region) after completion of PE on that day.
  * Subsequent days of treatment during PE: daily s.c. injection (in the abdominal region) following PE.
  * Treatment after PE period: daily s.c. injections for 30 days. If the underlying immunological disease was not resolved, treatment could be extended for a maximum of 4 additional 1-week periods (i.e., 28 days) and was to be accompanied by optimization of immunosuppression.
Period: Overall Treatment Period + Follow-up
Arm/Group | Caplacizumab | Placebo
Started | 72 | 73
Received Study Drug | 71 | 73
Completed | 58 | 50
Not Completed | 14 | 23
Not completed — Withdrawn by legal representative | 0 | 1
Not completed — Physician Decision | 2 | 4
Not completed — Non-compliance with study drug | 0 | 1
Not completed — Death | 1 | 3
Not completed — Adverse Event | 6 | 5
Not completed — Withdrawal by Subject | 4 | 5
Not completed — Lost to Follow-up | 0 | 1
Not completed — Diagnosed as non-TTP patient | 1 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrew treatment, agreed for ET visit | 0 | 1
Period: Double-blind (DB) Treatment Period
Arm/Group | Caplacizumab | Placebo
Started | 71 (One patient withdrew consent prior to first dosing and did not start the DB treatment period.) | 73
Completed | 68 | 65
Not Completed | 3 | 8
Period: Open-label (OL) Treatment Period
Arm/Group | Caplacizumab | Placebo
Started | 2 (2 patients on caplacizumab had a recurrence of TTP during the DB period and started OL treatment.) | 26 (26 patients on placebo had a recurrence of TTP during the DB period and started OL treatment.)
Completed | 2 | 22
Not Completed | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Caplacizumab: Caplacizumab 10 mg once daily
  Caplacizumab:
  * First day of treatment: 10 mg intravenous (i.v.) injection prior to PE followed by a 10 mg subcutaneous (s.c.) injection (in the abdominal region) after completion of PE on that day.
  * Subsequent days of treatment during PE: daily 10 mg s.c. injection (in the abdominal region) following PE.
  * Treatment after PE period: daily 10 mg s.c. injections for 30 days. If the underlying immunological disease was not resolved, treatment could be extended for a maximum of 4 additional 1-week periods (i.e., 28 days) and was to be accompanied by optimization of immunosuppression.
- Total: Total of all reporting groups
Arm/Group | Caplacizumab | Placebo | Total
Number analyzed (Participants) | 72 | 73 | 145
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 68 | 65 | 133
  >=65 years | 4 | 8 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.9 (13.46) | 47.3 (14.07) | 46.1 (13.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 51 | 100
  Male | 23 | 22 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 6
  Not Hispanic or Latino | 65 | 62 | 127
  Unknown or Not Reported | 3 | 9 | 12
Region of Enrollment [Count of Participants; unit: Participants]
  Hungary | 4 | 3 | 7
  United States | 10 | 22 | 32
  Czechia | 2 | 2 | 4
  United Kingdom | 13 | 8 | 21
  Switzerland | 1 | 0 | 1
  Spain | 8 | 6 | 14
  Canada | 7 | 6 | 13
  Austria | 3 | 1 | 4
  Netherlands | 1 | 0 | 1
  Turkey | 4 | 5 | 9
  Belgium | 5 | 3 | 8
  Italy | 6 | 4 | 10
  Israel | 4 | 2 | 6
  Australia | 1 | 2 | 3
  France | 3 | 9 | 12

OUTCOME MEASURES:

1. Primary Outcome: Time to Platelet Count Response
Description: Platelet count response was defined as initial platelet count ≥ 150,000/μL with subsequent stop of daily PE within 5 days. It refers to the first time both conditions, platelet count ≥ 150,000/μL and the stop of daily PE within 5 days, were met.
Time Frame: Only data from the DB daily PE period (median = 5 days) up to the cut-off were used. The cut-off point was defined by whichever occured first: 1) 45 days of daily PE after start of study drug, 2) stop of daily PE, 3) stop of study drug (median = 34 days)
Population: Intent-to-treat (ITT) population (for the respective study period, i.e., DB treatment period)
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Caplacizumab | Placebo
Number analyzed (Participants) | 71 | 73
days | 2.69 [1.89 to 2.83] | 2.88 [2.68 to 3.56]
Statistical Analysis 1: Comparison: Caplacizumab vs Placebo; Time to platelet count response in the caplacizumab arm and placebo arm was compared by conducting a two-sided stratified log-rank test based on a KM analysis, with severity of neurological involvement (according to the Glasgow coma scale [GCS] category, stratification factor used in randomization: ≤12 / 13-15) as stratification factor; Test type: Superiority; p = 0.0099, Log Rank — The resulting p-value was compared with a significance level of 5%
Statistical Analysis 2: Comparison: Caplacizumab vs Placebo; Time to platelet count response was analyzed using a Cox proportional hazards regression model with time to platelet count response as dependent variable, and treatment group and GCS category as independent variables. The hazard (or platelet count normalization rate) ratio from the Cox model was reported along with 95% CI; Test type: Superiority; Hazard Ratio (HR) = 1.55, 95% CI 2-sided [1.095 to 2.195] — The HR was estimated from a Cox proportional Hazards regression model

2. Secondary Outcome: Number and Percentage of Subjects With TTP-Related Death, Recurrence of TTP, or a Major Thromboembolic Event During the Study Drug Treatment Period
Description: Number and percentage of subjects with TTP-related death, a recurrence of TTP, or at least one treatment-emergent major thromboembolic event during the study drug treatment period (i.e., first key secondary endpoint).
Time Frame: The study drug treatment period, a median (min, max) of 36 (2, 82) days. For both treatment groups, only events that occurred prior to a switch to open-label caplacizumab were evaluated for this analysis.
Population: ITT Population (for the respective study period, i.e., overall treatment period)
Measure: Count of Participants; unit: Participants
Arm/Group | Caplacizumab | Placebo
Number analyzed (Participants) | 71 | 73
Participants | 9 | 36
Statistical Analysis 1: Comparison: Caplacizumab vs Placebo; A Cochran-Mantel-Haenszel (CMH) test was conducted with adjustment for GCS category (stratification factor used in randomization); Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — The resulting p-value was compared with a significance level of 5%

3. Secondary Outcome: Number and Percentage of Subjects With a Recurrence of TTP in the Overall Study Period
Description: Number and percentage of subjects with a recurrence of TTP during the Overall Study Period (i.e., including follow-up [FU]) (i.e., second key secondary endpoint).
Time Frame: The overall study period (covers both the overall treatment period and the follow-up period), a median (min, max) of 65 (2, 110) days.
Population: ITT Population (for the respective study period, i.e., overall study period)
Measure: Count of Participants; unit: Participants
Arm/Group | Caplacizumab | Placebo
Number analyzed (Participants) | 71 | 73
Participants | 9 | 28
Statistical Analysis 1: Comparison: Caplacizumab vs Placebo; A CMH test was conducted with adjustment for GCS category (stratification factor used in randomization); Test type: Superiority; p = 0.0004, Cochran-Mantel-Haenszel — The resulting p-value was compared with a significance level of 5%

4. Secondary Outcome: Number and Percentage of Subjects With Refractory Disease
Description: Number and percentage of subjects with refractory TTP, defined as absence of platelet count doubling after 4 days of standard treatment, and lactate dehydrogenase (LDH) > upper limit of normal (ULN) (i.e., third key secondary endpoint).
Time Frame: The study drug treatment period, a median (min, max) of 36 (2, 82) days.
Population: ITT Population (for the respective study period, i.e., overall treatment period)
Measure: Count of Participants; unit: Participants
Arm/Group | Caplacizumab | Placebo
Number analyzed (Participants) | 71 | 73
Participants | 0 | 3
Statistical Analysis 1: Comparison: Caplacizumab vs Placebo; A CMH test was conducted with adjustment for GCS category (stratification factor used in randomization); Test type: Superiority; p = 0.0572, Cochran-Mantel-Haenszel — The resulting p-value was compared with a significance level of 5%

5. Secondary Outcome: Time to Normalization of Organ Damage Marker Levels
Description: Time to first normalization of LDH, cardiac troponin I (cTnI) and serum creatinine was defined as: first time of LDH ≤ ULN and cTnI ≤ ULN and serum creatinine ≤ ULN - time of first i.v. loading dose of study drug after randomization + 1 minute. Subjects in either initial treatment group who switched to open-label caplacizumab before having reached the endpoint were censored at time of switch.
  Of note, the key secondary endpoints were hierarchically ordered to allow statistical testing for these endpoints at the same nominal significance level of 5% without adjustment, as long as the tests occurred in the pre-defined sequential order, and given that all null hypotheses tested for endpoints with a higher rank (including the primary endpoint) were rejected. No confirmatory testing was done for this fourth key secondary endpoint, as the statistical test was not significant for the proportion of subjects with refractory disease (i.e., the third key secondary endpoint).
Time Frame: Overall study period, a median (min, max) of 65 (2, 110) days. For both treatment groups, normalizations occurring during the open-label period were not evaluated in this analysis.
Population: ITT Population (for the respective study period, i.e., overall study period) with biomarker level data available
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Caplacizumab | Placebo
Number analyzed (Participants) | 65 | 66
days | 2.86 [1.93 to 3.86] | 3.36 [1.88 to 7.71]

6. Other Pre Specified Outcome: Number of Days of Plasma Exchange
Description: The number of days of PE during the overall study drug treatment period, including the number of days of PE during the open-label study drug treatment period. Data were analyzed according to the initial treatment allocation (both before and after switch to open-label caplacizumab).
Time Frame: Overall study drug treatment period, a median (min, max) of 36 (2, 82) days.
Population: ITT Population (for the respective study period, i.e., overall treatment period)
Measure: Mean (Standard Error); unit: days
Arm/Group | Caplacizumab | Placebo
Number analyzed (Participants) | 71 | 73
days | 5.8 (0.51) | 9.4 (0.81)

7. Other Pre Specified Outcome: Total Volume of Plasma Exchange
Description: The total volume of PE during the overall study drug treatment period, including the total volume of PE during the open-label study drug treatment period. Data were analyzed according to the initial treatment allocation (both before and after switch to open-label caplacizumab).
Time Frame: Overall study drug treatment period, a median (min, max) of 36 (2, 82) days.
Population: ITT Population (for the respective study period, i.e., overall treatment period)
Measure: Mean (Standard Error); unit: liter(s)
Arm/Group | Caplacizumab | Placebo
Number analyzed (Participants) | 71 | 73
liter(s) | 21.33 (1.619) | 35.93 (4.169)

8. Other Pre Specified Outcome: Number of Days in Intensive Care Unit
Description: The number of days in intensive care unit (ICU) during the overall study drug treatment period, including the number of days in ICU during the open-label study drug treatment period. Data were analyzed according to the initial treatment allocation (both before and after switch to open-label caplacizumab).
Time Frame: Overall study drug treatment period, a median (min, max) of 36 (2, 82) days.
Population: ITT Population (for the respective study period, i.e., overall treatment period)
Measure: Mean (Standard Error); unit: days
Arm/Group | Caplacizumab | Placebo
Number analyzed (Participants) | 71 | 73
days | 3.4 (0.40) | 9.7 (2.12)

9. Other Pre Specified Outcome: Number of Days in Hospital
Description: The number of days in hospital during the overall study drug treatment period, including the number of days in hospital during the open-label study drug treatment period. Data were analyzed according to the initial treatment allocation (both before and after switch to open-label caplacizumab).
Time Frame: Overall study drug treatment period, a median (min, max) of 36 (2, 82) days.
Population: ITT Population (for the respective study period, i.e., overall treatment period)
Measure: Mean (Standard Error); unit: days
Arm/Group | Caplacizumab | Placebo
Number analyzed (Participants) | 71 | 73
days | 9.9 (0.70) | 14.4 (1.22)

ADVERSE EVENTS:
Time Frame: From time of first study drug administration until the subject's study completion/discontinuation date, a median (min, max) of 65 (2, 110) days.
Description: Double-Blind Caplacizumab/Double-Blind placebo groups (subjects randomized to caplacizumab/placebo, respectively): adverse events (AEs) starting in DB or FU Periods for subjects with no OL Period. Only AEs starting in the DB Period for subjects with an OL Period.
  OL Caplacizumab group (all subjects with OL Period): AEs starting in the OL or FU Periods.
  The 3 subjects who died in the placebo group died during treatment and the subject who died in the caplacizumab group died during follow-up.
Groups:
- Double-blind Caplacizumab: Caplacizumab 10 mg once daily
- Double-blind Placebo: Placebo once daily
- Open-label Caplacizumab: In case an exacerbation during the 30-day treatment period or a relapse during the treatment extension period occurred (first exacerbation or relapse), subjects were to receive open label caplacizumab 10 mg daily together with re-initiation of daily PE and optimized immunosuppressive treatment. Caplacizumab treatment schedule and visit schedule were the same as for the initial study drug treatment period (covering daily PE [variable duration] and 30-day post-daily PE period) and the possible treatment extension period.
Arm/Group | Double-blind Caplacizumab | Double-blind Placebo | Open-label Caplacizumab
All-Cause Mortality (participants affected / at risk) | 1/71 | 3/73 | 0/28
Serious Adverse Events (participants affected / at risk) | 28/71 | 39/73 | 7/28
Other Adverse Events (participants affected / at risk) | 67/71 | 65/73 | 25/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-blind Caplacizumab (N=71) | Double-blind Placebo (N=73) | Open-label Caplacizumab (N=28)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal ischemia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebral ischemia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hemorrhagic transformation stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Rash erythematosus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 9 (9) | 29 (29) | 4 (4)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) — Verbatim term of serious adverse event (SAE) with fatal outcome: septic shock
Bacteremia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Device related sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 0 (0)
Subarachnoid hemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Arteriospasm coronary (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Hemorrhagic ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Gallbladder necrosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Serum sickness (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-blind Caplacizumab (N=71) | Double-blind Placebo (N=73) | Open-label Caplacizumab (N=28)
Catheter site hemorrhage (General disorders) | 5 (6) | 5 (5) | 8 (10)
Fatigue (General disorders) | 10 (10) | 6 (6) | 2 (2)
Pyrexia (General disorders) | 10 (12) | 6 (6) | 1 (1)
Oedema peripheral (General disorders) | 4 (4) | 7 (8) | 1 (2)
Asthenia (General disorders) | 2 (3) | 4 (4) | 2 (3)
Chest pain (General disorders) | 1 (1) | 5 (6) | 1 (1)
Catheter site pain (General disorders) | 1 (1) | 5 (5) | 0 (0)
Injection site pain (General disorders) | 1 (1) | 4 (4) | 1 (1)
Injection site hematoma (General disorders) | 1 (1) | 3 (4) | 2 (2)
Pain (General disorders) | 4 (7) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 1 (1) | 1 (1) | 2 (4)
Injection site pruritus (General disorders) | 2 (2) | 0 (0) | 2 (2)
Injection site reaction (General disorders) | 1 (1) | 0 (0) | 2 (2)
Face oedema (General disorders) | 0 (0) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 10 (12) | 7 (8) | 2 (2)
Gingival bleeding (Gastrointestinal disorders) | 12 (13) | 1 (1) | 4 (5)
Constipation (Gastrointestinal disorders) | 7 (7) | 5 (6) | 4 (6)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 5 (5) | 4 (7)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 4 (4) | 2 (4)
Vomiting (Gastrointestinal disorders) | 3 (3) | 4 (5) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 4 (8)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2)
Hematochezia (Gastrointestinal disorders) | 2 (5) | 0 (0) | 2 (2)
Lip hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 14 (18) | 6 (10) | 6 (6)
Dizziness (Nervous system disorders) | 7 (8) | 8 (8) | 2 (3)
Paresthesia (Nervous system disorders) | 8 (9) | 6 (6) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 12 (14) | 5 (8) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 5 (6) | 9 (11) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (6) | 6 (6) | 2 (4)
Petechiae (Skin and subcutaneous tissue disorders) | 4 (4) | 5 (5) | 3 (5)
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 21 (32) | 2 (2) | 5 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (10) | 2 (2) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 4 (4) | 6 (9) | 4 (8)
Urinary tract infection (Infections and infestations) | 4 (4) | 4 (4) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 4 (4) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (5) | 6 (7) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 (5) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 2 (3)
Hypokalemia (Metabolism and nutrition disorders) | 6 (6) | 14 (15) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (5) | 4 (4) | 1 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 5 (8) | 2 (3)
Insomnia (Psychiatric disorders) | 6 (7) | 8 (8) | 0 (0)
Anxiety (Psychiatric disorders) | 4 (4) | 6 (6) | 1 (1)
Agitation (Psychiatric disorders) | 5 (6) | 4 (4) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 5 (7) | 10 (24) | 2 (10)
Hypertension (Vascular disorders) | 4 (4) | 8 (8) | 1 (1)
Hematoma (Vascular disorders) | 3 (7) | 2 (2) | 2 (2)
Hypotension (Vascular disorders) | 4 (4) | 2 (3) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 4 (4) | 3 (5) | 1 (4)
Tachycardia (Cardiac disorders) | 2 (2) | 4 (4) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1) | 2 (2)
Hematuria (Renal and urinary disorders) | 5 (7) | 2 (2) | 2 (2)
Vaginal hemorrhage (Reproductive system and breast disorders) | 4 (5) | 2 (2) | 1 (1)
Vision blurred (Eye disorders) | 5 (6) | 5 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of any results from this study will be according to the principles of the Declaration of Helsinki, in particular point 30, and will require prior review and written agreement of the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2016-07-20): https://cdn.clinicaltrials.gov/large-docs/17/NCT02553317/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-14): https://cdn.clinicaltrials.gov/large-docs/17/NCT02553317/SAP_001.pdf